CLINICAL TRIAL: NCT02581293
Title: Effect of Visceral and Parietal Peritoneum Suturation on Postoperative Vital Signs
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, MERYEM Kurek EKEN, M.D, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 31/2015
Record Dates: First submitted 2015-09-16; First posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Only visceral peritoneum will be closed (Experimental): Group1: Only visceral peritoneum will be closed
  Interventions: Procedure: Group 1: Only visceral peritoneum will be closed
- Only parietal peritoneum will be closed (Experimental): Group 2: Only parietal peritoneum will be closed
  Interventions: Procedure: Group 2 : Only parietal peritoneum will be closed
- Both of them will be closed (Experimental): Group 3: Both of them will be closed
  Interventions: Procedure: Group 3 : Both of them will be closed
- None of them will be closed (Experimental): Group 4: None of them will be closed
  Interventions: Procedure: Group 4: None of them will be closed

INTERVENTIONS:
Procedure: Group 1: Only visceral peritoneum will be closed
  Arms: Only visceral peritoneum will be closed
Procedure: Group 2 : Only parietal peritoneum will be closed
  Arms: Only parietal peritoneum will be closed
Procedure: Group 3 : Both of them will be closed
  Arms: Both of them will be closed
Procedure: Group 4: None of them will be closed
  Arms: None of them will be closed

SUMMARY:
In this study the investigators want to asses the effect of peritonisation at c-section on postoperative vital signs which was thought to be an indirect finding secondary to increased sympathetic activity originated from pain caused by stretched peritoneum.

DETAILED DESCRIPTION:
At c-section subject will be randomised into four groups:

Group1: Only visceral peritoneum will be closed

Group 2: Only parietal peritoneum will be closed

Group 3: Both of them will be closed

Group 4: None of them will be closed

During the postoperative period all patients will undergo vital sign screening including urine output, blood pressure measurement, pulse rate and VAS score will be determined at post operative 6th hour and 24th hour.

ELIGIBILITY:
Inclusion Criteria:

* Women underwent uncomplicated c-section

Exclusion Criteria:

* Patient with systemic Diseases
* Pregnant with Obstetric complications
* Pregnant with two or more previous c-sections

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 132 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative vital sign (arterial tension) | First postoperative hour

CONTACTS AND LOCATIONS:
Overall Officials: Enis Özkaya, Assoc. Prof., Principal Investigator — Zeynep Kamil Education and Research Hospital Obstetric and Gynecology Department
Locations (1):
- Meryem Kurek EKEN, Istanbul, Üsküdar, Turkey (Türkiye)